CLINICAL TRIAL: NCT07209111
Title: A Phase 2, Open-Label, Multicenter, Tumor-agnostic Study of MK-1084 as Monotherapy and in Combination With Cetuximab, in Participants With KRAS G12C-Mutant, Advanced Solid Tumors (KANDLELIT-014)
Brief Title: A Clinical Study of Calderasib (MK-1084) in People With Advanced Solid Tumors (MK-1084-014)
Acronym: KANDLELIT-014
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1084-014; MK-1084-014 (Other: MSD); U1111-1320-8626 (Registry Identifier: UTN); 2025-521737-91-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neoplasm Malignant
Keywords: KRAS; NSCLC; CRC; Tumor-agnostic; Pan Tumor; KRAS G12C
MeSH Terms: conditions — Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Calderasib (Experimental): Participants will receive calderasib orally. Per protocol treatment of calderasib has no maximum number of cycles. Participants will be treated until any of the criteria for discontinuation of study intervention are met.
  Interventions: Drug: Calderasib
- Calderasib + Cetuximab (Experimental): Participants will receive calderasib orally. Participants will receive Cetuximab 500 mg/m^2 via intravenous (IV) infusion once every 2 weeks (Q2W). Per protocol treatment of calderasib and Cetuximab has no maximum number of cycles. Participants will be treated until any of the criteria for discontinuation of study intervention are met.
  Interventions: Drug: Calderasib; Biological: Cetuximab

INTERVENTIONS:
Drug: Calderasib — Oral administration
  Other Names: MK-1084
Biological: Cetuximab — Intravenous administration
  Arms: Calderasib + Cetuximab

SUMMARY:
Researchers want to learn if calderasib given alone or with cetuximab can treat certain advanced solid tumors in people with the KRAS G12C mutation.

The goals of this study are to learn:

* How many people have the cancer respond (get smaller or go away) to calderasib alone or with cetuximab and how these responses compare
* About the safety of calderasib alone or with cetuximab and if people tolerate the treatments.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has locally advanced unresectable or metastatic solid tumor malignancy other than colorectal cancer and has progressed on, or following, standard of care systemic treatment
* Has a tumor that demonstrates the presence of Kirsten rat sarcoma (KRAS) G12C mutation

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system metastases and/or carcinomatous meningitis and/or primary brain tumors
* Has active infection, other than those permitted per protocol, requiring systemic therapy
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2032-04-09 (Estimated); Study Completion 2032-04-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 76 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 76 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 76 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 76 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Duration of Response (DOR) | Up to approximately 76 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 76 months
  OS is defined as the time from randomization to the date of death due to any cause. OS will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- United States (4):
  - Greater Baltimore Medical Center ( Site 1104), Baltimore, Maryland
  - START Midwest ( Site 1103), Grand Rapids, Michigan
  - START Mountain Region ( Site 1106), West Valley City, Utah
  - Virginia Cancer Specialists ( Site 1102), Fairfax, Virginia
- Denmark (2):
  - Rigshospitalet ( Site 1403), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 1401), Odense, Region Syddanmark
- Universitätsklinikum Jena ( Site 1603), Jena, Thuringia, Germany
- Israel (3):
  - Emek Medical Center ( Site 1800), Afula
  - Hadassah Medical Center ( Site 1801), Jerusalem
  - Sourasky Medical Center ( Site 1802), Tel Aviv
- Italy (2):
  - Istituto Clinico Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1902), Rozzano, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1900), Milan
- Norway (2):
  - Haukeland universitetssykehus ( Site 2102), Bergen, Hordaland
  - Oslo universitetssykehus, Radiumhospitalet ( Site 2101), Oslo
- MTZ Clinical Research powered by Pratia ( Site 2205), Warsaw, Masovian Voivodeship, Poland
- South Korea (3):
  - Seoul National University Hospital ( Site 2301), Seoul
  - Asan Medical Center ( Site 2302), Seoul
  - Samsung Medical Center ( Site 2300), Seoul
- Spain (4):
  - Hospital Virgen de la Victoria ( Site 2403), Málaga, Malaga
  - Hospital Universitari Vall d Hebron ( Site 2401), Barcelona
  - Hospital Clinic de Barcelona ( Site 2402), Barcelona
  - Hospital Clinico San Carlos ( Site 2404), Madrid
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna ( Site 2501), Stockholm, Stockholm County
  - Sahlgrenska Universitetssjukhuset. ( Site 2502), Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/